CLINICAL TRIAL: NCT05511220
Title: Amplifying Treatment Response in Early Intervention 'Minimal Responders' With Autism Spectrum Disorder: A Virtual Parent-Coaching Intervention
Brief Title: Pivotal Response Intervention Minimal Responders Study
Acronym: PRIMeR
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: IWK Health Centre (Other)
Collaborators: Canadian Institutes of Health Research (CIHR) (Other Government)
Responsible Party: Principal Investigator, Dr. Isabel Smith, Professor; Joan & Jack Craig Chair in Autism Research, IWK Health Centre
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: 1027196
Record Dates: First submitted 2022-08-05; First posted 2022-08-22 (Actual); Last update posted 2022-08-22 (Actual); Status verified 2022-08

CONDITIONS: Autism Spectrum Disorder With Impaired Functional Language
Keywords: autism spectrum disorder; limited verbal ability; early intervention; parent-mediated intervention
MeSH Terms: conditions — Autism Spectrum Disorder | interventions — DNA Primers

STUDY DESIGN:
Intervention Model Description: Hierarchical modelling will be used to examine aggregated data from multiple single case experimental design (SCED) series (n = 5 per series), with participants randomized to 1 of 2 treatment conditions. Target is 4 SCED series per treatment condition, therefore N of 20 per condition. See Jaksic et al. (2018) for information on this method.
Who Masked: Outcomes Assessor
Masking Description: Primary outcome will be coded by raters who are trained to 80% reliability on a coding scheme with operational definitions, and naive to treatment condition and study phase
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- PRIMeR (Experimental): Virtual parent coaching in use of a novel intervention consisting of Social Routines and Reciprocal Imitation Training strategies
  Interventions: Behavioral: PRIMeR
- PRT (Active Comparator): Virtual parent coaching in use of Pivotal Response Treatment strategies
  Interventions: Behavioral: PRT

INTERVENTIONS:
Behavioral: PRIMeR — Virtual PRIMeR intervention consists of coaching parents to use strategies derived from Social Routines (to boost positive affect) and Reciprocal Imitation Training (to boost toy play)
  Other Names: Social Routines; Reciprocal Imitation Training
  Arms: PRIMeR
Behavioral: PRT — Virtual PRT intervention consists of coaching parents to use key PRT strategies to enhance children's communication skills
  Other Names: Pivotal Response Treatment
  Arms: PRT

SUMMARY:
Early intervention (EI) using naturalistic behavioural methods have shown benefits for the development of communication and other skills for young children with autism spectrum disorder. The publicly funded autism EI program in Nova Scotia (NS) is based on such a method, Pivotal Response Treatment (PRT), and pre-post studies indicate benefits for children and families. However, not all children benefit equally. In this study, the investigators test the efficacy of a brief parent-mediated intervention designed to prime responsivity to PRT in children with a minimal responder profile derived from previous studies of the PRT-based EI program.

DETAILED DESCRIPTION:
Investigators will enroll preschoolers with the minimal responder profile who are scheduled to begin the PRT-based public EI program. Consenting parents will be offered a virtual intervention in which they will be randomized to 1 of 2 arms to receive coaching in either (a) PRIMeR intervention, designed to target areas of weakness in the minimal responder profile, or (b) PRT, the treatment model used in the EI program. Coaching will take place on a virtual (video-conferencing) platform. Each child's progress on treatment targets will be assessed in a single case experimental design (SCED) using data from blind-coded video-recordings of parent-child play episodes using a standard set of toys. Overall study effects will be based on aggregated data for an anticipated n of 20 participants assigned to each arm (4 SCED series with 5 participants each contributing to each arm). The primary outcome is gains in children's social initiations (video-coded); the secondary outcome is gains in children's communication levels (multi-method assessment). Mixed methods will be used to evaluate aspects of parents' experiences,

ELIGIBILITY:
Inclusion Criteria:

1. upcoming enrollment in NS EI program for preschoolers with autism spectrum disorder (ASD), based on confirmed or provisional ASD diagnosis by a qualified clinician
2. significant delay in cognitive abilities (assessed formally by psychologist or estimated by psychologist or developmental pediatrician at time of diagnosis)
3. current spontaneous functional use of ≤ 10 words (clinician's observations; parent report using MacArthur-Bates Communicative Development Inventory - Words & Gestures (CDI-WG)
4. limited use of toys / objects (clinician's impression or parent's report with no contrary observation by clinician)
5. low levels of expressed positive affect (smiles, laughter) or limited positive and high negative affect (clinician's impression or parent's report with no contrary observation by clinician)

Exclusion Criteria:

1. Severe sensory or motor impairment in child
2. Parent unable to complete consent process (and receive coaching) in English

Ages: 3 Years to 5 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 40 (Estimated)
Dates: Start 2022-07-12 (Actual); Primary Completion 2024-10 (Estimated); Study Completion 2025-03-30 (Estimated)

PRIMARY OUTCOMES:
Social initiations | Assessed at baseline, entry to EI program, and after 6 months of EI program
  Change in frequency of child's social initiations toward parent, blind-coded from video sample

SECONDARY OUTCOMES:
Communication | Assessed at baseline, entry to EI program, and after 6 months of EI program
  Change in level of communication derived from Assessment of Phase of Preschool Language (APPL)

CONTACTS AND LOCATIONS:
Overall Officials: Isabel M Smith, PhD, Principal Investigator — IWK Health Centre and Dalhousie University
Locations (1):
- IWK Health Centre, Halifax, Nova Scotia, Canada

IPD SHARING:
Plan to Share IPD: No